CLINICAL TRIAL: NCT00878956
Title: A Phase IIb Multiple Blind Randomized Controlled Trial of Sodium Bicarbonate in Cardiac Surgery at High-risk of Acute Kidney Injury
Brief Title: Bicarbonate in Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of ICU Research, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2007/02808
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Acute Kidney Injury
Keywords: Cardiac surgery; Cardiopulmonary bypass; Oxidative stress; Acute renal dysfunction; Sodium bicarbonate
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium bicarbonate at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Interventions: Drug: Sodium Bicarbonate
- 2 (Placebo Comparator): In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium chloride at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Sodium Bicarbonate — In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium bicarbonate at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Arms: 1
Drug: Sodium Chloride — In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium chloride at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Arms: 2

SUMMARY:
With over one million operations a year, cardiac surgery with cardiopulmonary bypass is one of the most common major surgical procedures worldwide (1). Acute kidney injury is a common and serious postoperative complication of cardiopulmonary bypass and may affect 25% to 50% of patients (2-4). Acute kidney injury carries significant costs (4) and is independently associated with increased morbidity and mortality (2,3). Even minimal increments in plasma creatinine are associated with an increase in mortality (5,6).

Multiple causes of cardiopulmonary bypass-associated acute kidney injury have been proposed, including ischemia-reperfusion, generation of reactive oxygen species, hemolysis and activation of inflammatory pathways (7-10). To date, no simple, safe and effective intervention to prevent cardiopulmonary bypass-associated acute kidney injury in a broad patient population has been found (11-14).

Urinary acidity may enhance the generation and toxicity of reactive oxygen species induced by cardiopulmonary bypass (10,15). Activation of complement during cardiac surgery (16) may also participate in kidney injury. Urinary alkalinization may protect from kidney injury induced by oxidant substances, iron-mediated free radical pathways, complement activation and tubular hemoglobin cast formation (9,17,18). Of note, increasing urinary pH - in combination with N-acetylcysteine (19,20) or without (21) - has recently been reported to attenuate acute kidney injury in patients undergoing contrast-media infusion.

In a pilot double-blind, randomized controlled trial the investigators found sodium bicarbonate to be efficacious, safe, inexpensive and easy to administer. These findings now need to be confirmed or refuted by further clinical investigations in other geographic and institutional settings.

Accordingly, the investigators hypothesized that urinary alkalinization might protect kidney function in patients at increased risk of acute kidney injury undergoing cardiopulmonary bypass needs to be confirmed in an international multicenter, double-blind, randomized controlled trial of intravenous sodium bicarbonate.

DETAILED DESCRIPTION:
Renal impairment following cardiopulmonary bypass is common. While most of these patients do not require either short or long term renal replacement, the mortality of patients with acute renal failure is substantially greater than those who do not develop renal dysfunction.

In a pilot double-blind, randomized controlled trial we found sodium bicarbonate to be efficacious, safe, inexpensive and easy to administer. These findings now need to be confirmed or refuted by further clinical investigations in other geographic and institutional settings.

There is evidence that sodium bicarbonate affects the cardiovascular, respiratory and immune systems and may be of benefit to patients undergoing cardiac surgery.

Study Design - overview and rationale

Patients will be randomised to receive sodium bicarbonate from the induction of anaesthesia until 24 hours postoperatively, or a placebo (sodium chloride).

Serum creatinine is the most commonly used clinical indicator of renal function along with urine output. Both will be measured for several days postoperatively - the time period during which renal impairment is most likely to develop.

Randomisation The randomisation will be based on random numbers generated by computer. Once consent is obtained, the allocation of either treatment with sodium bicarbonate or placebo will be organised by an independent person (clinical trials pharmacist) who will dispense the coded and blinded infusion bags (shrink-wrapped in extra black plastic bags). This will be delivered to the anaesthetic staff looking after the patient in theatre, and the ICU nurse caring for the patient postoperatively.

20 ml samples of heparinised blood and urine will be taken from the arterial line or urine catheter. Samples will be taken immediately after the preoperative insertion of the arterial/urine catheter, at 6, 24, 48, 72, 96 and 120 hours after commencement of cardiopulmonary bypass. Immediately following collection, the preoperative, 6 and 24 hour blood and urine will be centrifuged at low speed to separate the plasma from the cellular components. Urine and plasma will be stored in aliquots at -70 degrees prior to batch analysis.

The following variables will be obtained:

Code for patient, gender and age. Date and time of admission to ICU Operative procedure and date and time on and off cardiopulmonary bypass Preoperative assessment of left ventricular function, Comorbidities, Pre-, intra- and post-operative medication, Markers of renal function as described above, Doses of frusemide administered (or rate of frusemide infusion) Use of inotropes or vasopressors Cardiac output whenever measured for clinical purposes in the first 24 hours postoperatively Requirement of renal replacement therapy Urine output in each 6 hour period during the presence of urine catheter Acid base status and electrolytes at baseline, 6 and 24 hours after commencement of cardiopulmonary bypass, Time of intubation and extubation, Date and time of arrival on and discharge from ICU and hospital, death Resources required The principle of the study has been discussed with the involved cardiac anaesthetists, cardiac surgeons, intensivists and intensive care nurses, who have offered their co-operation. ICU research nurse to allocate patients and collect clinical data. Pharmacy will be required to prepare drug and placebo infusion bags. Clinical pathology will be required to perform 24 hour creatinine clearance estimation (in addition to those tests clinically indicated) Protocol violations All protocol violations will be recorded. It will then be decided whether the nature of such violation had been such that the patient should be excluded from primary data analysis. Such evaluation will be blinded to treatment.

Withdrawal

The treating clinician will have the right to withdraw the patient from the study if he or she believes that continued participation is jeopardising the patient's well being.

Ethical Issues

Sodium bicarbonate used in this study is considered to be very safe as has been demonstrated by its widespread clinical use in the management of critically ill patients with metabolic acidosis. We consider the potential benefit of this treatment theoretically significant. Given the balance of benefits and risks, we consider it ethical to proceed and seek informed consent.

Indemnity

This is an investigator-initiated study and, accordingly, no commercial sponsor's indemnity has been provided.

Informed consent will be obtained from the patient prior to the operation by one of the investigators or the ICU research nurse. The clinical care of a patient who does not consent for any reason will not be affected.

ELIGIBILITY:
Inclusion Criteria:

* Age above 70 years
* Pre-existing renal impairment (preoperative plasma creatinine concentration > 1.4 mg/dL
* New York Heart Association class III/IV or impaired left ventricular function (left ventricular ejection fraction < 50%)
* Valvular surgery or concomitant valvular and coronary artery bypass graft surgery
* Redo cardiac surgery
* Insulin-dependent diabetes mellitus

Exclusion Criteria:

* End stage renal disease (plasma creatinine concentration > 3.4 mg/dL)
* Emergency cardiac surgery
* Planned off-pump cardiac surgery
* Known blood-borne infectious disease
* Chronic inflammatory disease on immunosuppression
* Chronic moderate to high dose corticosteroid therapy (> 10 mg/d prednisone or equivalent)
* Enrolled in conflicting research study
* Age < 18 years

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 427 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine greater than 25% or 44 mmol/L (0.5 mg/dL) postoperative increase in serum creatinine after adjustment for relevant baseline variables | within first five postoperative days

SECONDARY OUTCOMES:
Mean changes in serum creatinine after adjustment for relevant baseline variables | within first five postoperative days
mean changes in serum cystatin C after adjustment for relevant baseline variables | within first five postoperative days
mean changes in urinary neutrophil gelatinase-associated lipocalin (NGAL)after adjustment for relevant baseline variables | within first five postoperative days
Duration of ventilation | Until time of extubation from mechanical ventilation
Proportion of patients developing any of the RIFLE criteria: R, I or F | within first five postoperative days
Incidence of post-operative atrial fibrillation | within first five postoperative days
Duration of stay in the intensive care unit (ICU) | from admission to the ICU
Duration of stay in hospital | from admission to discharge from hospital
90-day mortality | during 90 days postoperatively
Change in electrolyte status from baseline to peak | within first 24-48hrs postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Principal Investigator — Austin Hospital, Melbourne Australia; Frank van Haren, MD, Study Chair — Waikato Hospital, Hamilton, New Zealand; Shay McGuinness, MB ChB, FRCA, FANZCA, Study Chair — Auckland City Hospital
Locations (4):
- Australia (2):
  - Austin Hospital, Melbourne, Victoria
  - Warringal Private Hospital, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton